CLINICAL TRIAL: NCT04800172
Title: The Possible Effects of Roflumilast on Obesity Related Disorders
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sara Mohammed Zayed, Pharm D, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 34538/3/21
Record Dates: First submitted 2021-03-11; First posted 2021-03-16 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Obesity; PreDiabetes
MeSH Terms: conditions — Obesity; Prediabetic State | interventions — Roflumilast

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: double-blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Roflumilast arm (Active Comparator)
  Interventions: Drug: Roflumilast
- Placebo arm (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Roflumilast — administration of roflumilast 500 mcg tablet once daily for 3 months.
  Arms: Roflumilast arm
Drug: placebo — administration of placebo tablet once daily for 3 months.
  Arms: Placebo arm

SUMMARY:
Evaluation of the possible effects of roflumilast on weight, glucose and lipid metabolism, insulin resistance, oxidative stress and inflammatory process in prediabetic obese subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Prediabetic patients (fasting blood glucose between 100 mg/dl and 125 mg/dl or HbA1C within the range 5.7% and 6.4%).
2. Obese subjects (BMI ≥30 kg/m2 and <40 kg/m2).

Exclusion Criteria:

1. Patients with morbid obesity (BMI > 40 kg/m2).
2. Patients already on weight lowering agents or weight loss program.
3. History or current diagnosis of major depressive disorder or other psychiatric disorders that in the opinion of the investigator would make participation unsafe for the participant.
4. Moderate to severe liver disease (Child-Pugh B or C), renal disease, thyroid disease, cardiovascular disease, peripheral vascular disease or coagulopathy.
5. Women will be excluded from our study if they are pregnant, breastfeeding, currently on contraceptive pills or if they plan to become pregnant prior to the end of the study.
6. Patients on medications that can interfere with glucose or lipid metabolism (e.g. hypoglycemic agents, corticosteroids, anti-hyperlipidemics, non-selective β-blockers thiazides, etc.) and subjects with organic causes of obesity.
7. Diabetic patients and patients with any inflammatory disease.
8. Smokers.
9. Patients on cytochrome P450 inducers (e.g. rifampicin, phenobarbital, carbamazepine, phenytoin, etc.)

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Change in patients body weight | baseline and 3 months later
  substracting pre-treatment from post-treatment values.
Change in blood glucose | baseline and 3 months later
  using glucose oxidase method for assessment of blood glucose and substracting pre-treatment from post-treatment values.
Change in plasma insulin level | baseline and 3 months later
  substracting pre-treatment from post-treatment values of plasma insulin.
Change in HOMA-IR index | baseline and 3 months later
  HOMA-IR will be calculated for all patients at baseline and 3 months later.
Change in blood lipid levels | baseline and 3 months later
  blood lipid levels will be measured at baseline and 3 months after treatment including total cholesterol, triglycerides, HDL-C and LDL-C.

SECONDARY OUTCOMES:
Changes in TNF-alfa serum level | baseline and 3 months later
  substracting pre-treatment from post-treatment values of TNF-alfa.
Changes in malondialdehyde serum level (MDA) | baseline and 3 months later
  substracting pre-treatment from post-treatment values of MDA.

CONTACTS AND LOCATIONS:
Overall Officials: Sara M Zayed, Principal Investigator — Tanta University
Locations (1):
- Sara Mohammad Zayed, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No
Data of outcomes and other research but not personal data are intended to be published in application to scientific journals